CLINICAL TRIAL: NCT03328390
Title: Analgesia for Laparotomy in Cancer Patients:Ultrasound-guided Quadratus Lumborum Block Versus Transversus Abdominis Plane Block
Brief Title: Analgesia for Laparotomy in Cancer Patients: Quadratus Lumborum Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alaa Mazy (Other)
Responsible Party: Sponsor-Investigator, Alaa Mazy, Associate professor of anesthesia and surgical intensive care, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS/15.12.97
Record Dates: First submitted 2017-10-28; First posted 2017-11-01 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Sensitivity Training Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus lumborum block Group (Experimental): ultrasound guided
  Interventions: Other: Quadratus lumborum block
- Transversus abdominis plane block Group (Active Comparator): ultrasound guided
  Interventions: Other: Transversus abdominis plane block

INTERVENTIONS:
Other: Quadratus lumborum block — 15 ml of 0.5% isobaric bupivacaine + 10 ml saline + 50 micro gram dexmedetomidine + epinephrine (1:100,000) for each side.
  Other Names: Group Q
  Arms: Quadratus lumborum block Group
Other: Transversus abdominis plane block — 15 ml of 0.5% isobaric bupivacaine + 10 ml of saline + 50 micro gram dexmedetomidine + epinephrine (1:100,000) for each side.
  Other Names: Group T
  Arms: Transversus abdominis plane block Group

SUMMARY:
Regional anesthesia of the abdomen significantly reduce postoperative pain, spare the systemic opioids and decrease postoperative nausea and vomiting. Multiple regional techniques can be performed at the neuro-axis (epidural), the nerve root (paravertebral) and the peripheral nerve (transversus abdominis plane).

Quadratus lumborum (QL) block is an addition into the league of truncal nerve block techniques that has been found to provide analgesia for abdominal surgeries. Several case reports have shown that local anesthetic injection around the quadratus lumborum muscle is effective in providing pain relief after various abdominal operations and in patients with chronic pain.

The study hypothesis is that quadratus lumborum block in single shot may be more superior to transversus abdominus plane block as regard intra-operative and the post-operative analgesia.

DETAILED DESCRIPTION:
This is a prospective randomized controlled study conducted at Oncology Center-Mansoura University.

102 patients were randomly allocated by closed envelope method into 2 equal groups:

* Quadratus lumborum block Group (Q) (n= 51): patients received 15 ml of 0.5% isobaric bupivacaine + 10 ml saline + 50 ug dexmedetomidine + epinephrine (1:100,000) for each side.
* Transversus abdominis plane Group (T) (n= 51): patients received 15 ml of 0.5% isobaric bupivacaine + 10 ml of saline + 50 ug dexmedetomidine + epinephrine (1:100,000) for each side.

All blocks were performed after induction of general anesthesia and approximately 15 min before the skin incision.

* Technique of ultrasound guided quadratus lumborum Block: patient lie in lateral position to obtain appropriate view of quadratus lumborum and transversus abdominins plane extension of lateral abdominal muscles. In this approach, a high-frequency linear transducer (7-12 MHZ) attached to ultrasound machine was placed in anterior axillary line to visualize the typical triple abdominal layers. At the junction of the tapered ends of abdominal muscles and quadratus lumborum, a 21 G cannula needle was inserted in plane and confirmed its position by injecting saline. Under ultrasound guidance, saline separating thoracolumbar fascia from muscle is observed then local anesthetic is injected.
* Technique of ultrasound guided Transversus abdominis plane Block: Patient lie in supine position and high-frequency linear transducer (7-12 MHZ) attached to ultrasound machine placed in anterior axillary line between costal margin and iliac crest to visualize the typical triple abdominal layers. A 21 G cannula needle is then moved forward from an anteromedial position in a posterior and lateral direction using an in-plane technique with the entry point in the skin being separated from the probe in order to improve needle visibility in the long axis. The needle tip is inserted between transversus abdominis muscle and internal oblique muscle then local anesthetic is injected to produce separation between the two muscle.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for open abdominal cancer surgery.
* American Society of Anesthesiologists physical status grade I and grade II.

Exclusion Criteria:

1. Patient refusal. 2. Neuromuscular diseases (as myopathies, myasthenia gravies, …...) 3. Hematological diseases, bleeding or coagulation abnormality. 4. Psychiatric diseases. 5. Local skin infection and sepsis at site of the block. 6. Known intolerance to the study drugs. 7. Body Mass Index > 40 Kg/m2.

-

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
The total dose of morphine consumption | postoperative: in the first 24-hour
  milligram

SECONDARY OUTCOMES:
the time to the first analgesic requirement | postoperative: in the first 24-hour
  hours
pain intensity by visual analogue scale (VAS) | postoperatively, at 0, 2, 4, 8, 16 and 24 hours
  0-10 point visual analogue scale. 0 is no pain, 10 the worst pain.
sedation score by Modified Ramsay sedation score | postoperative, at 0, 2, 4, 8, 16 and 24 hours
  1-6 scale, 1. Anxious, agitated, restless. 2. Awake, but tranquil and cooperative. 3. Responsive to commands only.
  4. Brisk response to light glabellar tap or loud auditory stimulus. 5. Sluggish response to light glabellar tap or loud auditory stimulus.
  6. No response to light glabellar tap or loud auditory stimulus.
postoperative nausea, vomiting | postoperative in the first 24 hours
  percent
Mean blood pressure | intraoperatively every 30 minutes, then at 0, 2, 4, 8,16 and 24 hours postoperatively.
  millimeter mercury
Heart rate | intraoperatively every 30 minutes, then at 0, 2, 4, 8,16 and 24 hours postoperatively.
  beat/minute

CONTACTS AND LOCATIONS:
Locations (1):
- Oncolgy Center, Mansoura University,, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after publication
Supporting Information: SAP, CSR
Time Frame: no limit